CLINICAL TRIAL: NCT05172830
Title: Hellenic Registry of Subjects Receiving the Ovation Alto™ Abdominal Stent Graft System
Brief Title: Hellenic Registry of Ovation Alto™ Abdominal Stent Graft System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Patras (Other); University Hospital of Crete (Other); University Hospital, Alexandroupolis (Other)
Responsible Party: Principal Investigator, Konstantinos Spanos, Principal Investigator, Larissa University Hospital
Other Study IDs: 986152150
Record Dates: First submitted 2021-11-15; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: EVAR; Endovascular aneurysm repair; Ovation Alto
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group/Cohort: Ovation Alto™ Abdominal Stent Graft System Eligible patients must meet all of the inclusion criteria and none of the exclusion criteria.
  Interventions: Device: Ovation Alto™ Abdominal Stent Graft System

INTERVENTIONS:
Device: Ovation Alto™ Abdominal Stent Graft System — Single occurrence permanent implantation of AAA device

SUMMARY:
This is a Hellenic Registry including both retrospective and prospective subjects receiving the Ovation Alto™ Abdominal Stent Graft System ("Ovation Alto™ Abdominal Stent Graft System Post-Market Study") in the treatment of abdominal aortic aneurysms (AAA). The Ovation Alto™ Hellenic Registry is intended to expand the clinical knowledge base by collecting data on subjects treated with the Ovation Alto™ Abdominal Stent Graft System in actual clinical practice during the first post-operative year.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Both IFU and non-adherence to IFU
* Subject intends to electively receive the Ovation Alto™ Abdominal Stent Graft System
* Subject has the ability and willingness to comply with all follow-up exams as indicated in clinical investigation plan

Exclusion Criteria:

* Subject's current participation in a concurrent randomized control trial (RCT) or investigational device/drug study which could confound study results.
* Life expectancy less than 1 year
* Pregnancy
* Subjects with poor renal function as indicated by a serum creatinine > 2.5mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated electively with Ovation Alto™ Abdominal Stent Graft System for Endovascular Aneurysm Repair
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 12 months
  Treatment success is defined as technical success, freedom from type I and III endoleaks at 12 months, freedom from stent graft migration > 10m at 12 months compared to 1 month baseline, freedom from AAA enlargement >5mm at 12 months (compared to 1-month baseline, freedom from AAA rupture through 12 months, freedom from conversion to open repair through 12 months, stent graft stenosis, occlusion or kink requiring secondary intervention through 12 months, thromboembolic event attributable to stent graft requiring secondary intervention through 12 months, stent fracture requiring secondary intervention through 12 months.

SECONDARY OUTCOMES:
Number and Classification of Endoleaks | 1 and 12 months
  Endoleak type Ia and Ib and III
Stent Graft Migration | 1 and 12 months
  Any proximal caudal Stent Graft Migration >10mm
Abdominal aortic aneurysm sac enlargement | 1 and 12 months
  Any sac enlargement > 5mm
Aortic neck alteration | 1 and 12 months
  Any neck diameter increase at supra-renal part of the aorta (at 0mm, 10mm and 20mm above the highest renal artery), and infra-renal part of the aorta (at 0mm, 7mm, and 15mm below the lowest renal artery). Measurements of the aortic neck angulation will also be included
Freedom from abdominal aortic aneurysm rupture | 1 and 12 months
  Recording of any abdominal aortic aneurysm rupture that takes place during the follow up after the procedure in order to assess freedom from this adverse event
Number of Secondary Interventions | 1 and 12 months
  Any secondary intervention stent-graft related including: proximal extension with a balloon expandable covered stent; stent graft extension distally to common iliac arteries; use of onyx for Endoleak Ia; bare metal stent in external iliac arteries
AAA-related mortality | 1 and 12 months
  Any aneurysm related mortality
Device-related Adverse Events (AEs) | 1 and 12 months
  Device-related Adverse Events: loss of latency, stent fracture, migration, Endoleak type I and III
Major adverse events | 1 and 12 months
  Including death, myocardial infarction, stroke, chronic renal disease, stent graft infection, amputation
Adherence to instruction for use | 12 months
  Recording of patients in terms of adherence to instructions for use according to the device manual

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Larisssa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No